CLINICAL TRIAL: NCT03831893
Title: Evaluation of Potentially Bioactive Foods With Respect to Effects on Metabolic Test Markers and Cognitive Variables
Brief Title: Metabolic Effects of Nopal in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate Professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-00980
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): A food product similar to the test products but without nopal
  Interventions: Other: control
- Nopal food product 1 (Experimental): Food product with Nopal
  Interventions: Other: Nopal food product 1
- Nopal food product 2 (Experimental): Food product with Nopal
  Interventions: Other: Nopal food product 2

INTERVENTIONS:
Other: Nopal food product 1 — Dried Nopal incorporated in a food product
  Arms: Nopal food product 1
Other: Nopal food product 2 — Dried Nopal incorporated in a food product
  Arms: Nopal food product 2
Other: control — Food Product without nopal
  Arms: Control

SUMMARY:
The overall goal is to increase the knowledge that can be used for the development of food products with anti-diabetic properties, with the purpose to facilitate healthier food choices for people. More specifically the purpose of this study is to evaluate effects on metabolic test markers of Nopal (Opuntia) in healthy humans.

DETAILED DESCRIPTION:
The study include three visits at the research unit. At two of the visits the test subjects consume nopal in different doses. At one visit the subjects will consume a reference product. The intervention products are consumed at breakfast (at 8.00) and metabolic effects are investigated 3 hours postprandially. Consumption of the intervention products is separated by a one week washout period.

ELIGIBILITY:
Inclusion Criteria:

Healthy men and women (non-smokers), BMI 18,5-30 kg/m2, and with no known metabolic disorders or food allergies will be recruited to the studies. The test subjects should consume a normal diet in accordance with the Nordic Nutrition Recommendations.

Exclusion Criteria:

Fasting blood glucose >6.1 mmol/L. Metabolic diseases or conditions. Food allergies or gastro- intestinal conditions. Consumption of probiotics, antibiotics or other drugs..

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Blood glucose tolerance | 3 hours after breakfast (measurements at fasting, at 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min and 180 min. Area under the curve is calculated and used in the statistical evaluations)
  Repeated blood glucose determinations in the postprandial period after breakfast. The area under the curve, using incremental changes from baseline, are used in the statistical evaluation to determine glucose tolerance.

SECONDARY OUTCOMES:
subjective appetite sensations | 3 hours after breakfast (measurements at fasting, at 30 min, 60 min, 90 min, 120 min, 150 min and 180 min. Area under the curve is calculated and used in the statistical evaluations)
  changes in subjective appetite sensations will be registered in the postprandial period at breakfast, using 0 - 100 mm visual analogue scales (VAS scale). The two end points of the scales (i.e. 0 mm and 100 mm) represent the minimum and maximum, respectively, agreement with a appetite sensation. The hunger sensations to measure are: hunger, satiety and desire to eat.The area under the curve are used in the statistical evaluation to determine
Mood | 3 hours after breakfast (measurements at fasting, at 30 min, 60 min, 90 min, 120 min, 150 min and 180 min. Mean values are calculated and used in the statistical evaluations)
  Changes in mood parameters (valence and activity) will be registered in the postprandial period after breakfast.The mood measurements will be assessed using the Swedish Core Affect Scale which included three self-reporting rating scales for evaluating valence (unpleasantness-pleasantness) and for activation (quietness-excitement), respectively. The subjective mood ratings are registered using 0 mm-100 mm VAS. The two end points of the scales (i.e. 0 mm and 100 mm) represent the minimum and maximum, respectively, agreement with a sensation to be rated.The valence rating is assessed by obtaining a mean rating of three scales graded from displeased-pleased, sad-glad and depressed-happy, respectively, and the rating of activation is assessed by obtaining a mean rating of three scales graded from sleepy-awake, passive-active and dull-peppy, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Food Technology, engineering and Nutrition, LTH, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No